CLINICAL TRIAL: NCT02604524
Title: Reducing Risks and Improving Glucose Control During Extended Exercise in Youth With T1DM: The AP Ski Camp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Chernavvsky, MD, CRC (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); DexCom, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Daniel Chernavvsky, MD, CRC, Principal Investigator, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18529; DP3DK106826-01 (NIH)
Record Dates: First submitted 2015-11-06; First posted 2015-11-13 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2017-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus (T1DM); Artificial Pancreas (AP); Sensor-Augmented Pump (SAP) Therapy; Closed Loop Control; Insulin Pump; Continuous Glucose Monitor (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Lymphoproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed-Loop Control (CLC) System (Experimental): Subjects will use the Closed-Loop Control system in an attempt to maintain blood glucose in a certain range during the day and at night during the trial.
  Interventions: Device: Closed-Loop Control
- Sensor Augmented Pump Therapy Group (Placebo Comparator): Subjects will manage their own glucose levels during the trial.
  Interventions: Other: Sensor Augmented Pump Therapy

INTERVENTIONS:
Device: Closed-Loop Control — Subjects will use the CLC during 5 nights/6 days at a ski camp.
  Other Names: CLC
  Arms: Closed-Loop Control (CLC) System
Other: Sensor Augmented Pump Therapy — Subjects using their personal pumps with study CGM.
  Other Names: SAP
  Arms: Sensor Augmented Pump Therapy Group

SUMMARY:
The biggest challenges for glycemic control during the day time involve meals and exercise variations, which are impacted by age, fitness level, duration, intensity and history of exercise. Meal variability has the benefit that meals are typically announced and quantified. Glucose control around exercise, on the other hand, is more complicated if the patient doesn't announce a change in activity level.

DETAILED DESCRIPTION:
The object of this study is to evaluate the Closed-Loop Control (CLC) in an environment where muscle glycogen is systematically depleted, glucose uptake systematically increased, and meal sizes are naturally larger than normal: a week of camp at high altitude, with the concomitant variable of oxygen consumption that this environment involves; during the winter, that will expose and challenge the different components of the system during cold temperatures, and with twice daily practice of physical activity designed to deplete glycogen reserves such as skiing.

This proposal aims to demonstrate the superiority of the CLC, also known as Artificial Pancreas (AP), compared to the state-of-the art system available on the market: Sensor-augmented pump (SAP). This system has shown to diminish hypoglycemic events by setting the alarms on the continues glucose monitor (CGM) and taken action, such as performing self-monitoring blood glucose (SMBG) and treating if it is confirm to be low.

ELIGIBILITY:
Inclusion Criteria: To be eligible for the study, a subject must meet the following:

1. Criteria for documented hyperglycemia (at least 1 must be met):

   * Clinical diagnosis of type 1 diabetes (C-peptide levels and antibody determinations are not required)
   * The diagnosis of type 1 diabetes is based on the investigator's judgment
2. Criteria for requiring insulin at diagnosis (both criteria must be met):

   * Daily insulin therapy for ≥ 12 months
   * Insulin pump therapy for ≥ 3 months
3. Age 10 - 25 years
4. Avoidance of acetaminophen-containing medications (i.e. Tylenol) while wearing the continuous glucose monitor.
5. Willingness to wear a continuous glucose sensor and physiological monitor for the duration of the study
6. Female subjects who are sexually active must be on acceptable method of contraception (e.g. oral contraceptive pill, diaphragm, IUD)

Exclusion Criteria: The presence of any of the following is an exclusion for the study:

1. Diabetic ketoacidosis in the past 6 months
2. Hypoglycemic seizure or loss of consciousness in the past 6 months
3. History of seizure disorder (except for hypoglycemic seizure)
4. History of any heart disease including coronary artery disease, heart failure, or arrhythmias
5. History of altitude sickness
6. Chronic pulmonary conditions that could impair oxygenation
7. Cystic fibrosis
8. Current use of oral glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
9. History of ongoing renal disease (other than microalbuminuria).
10. Subjects requiring intermediate or long-acting insulin (such as NPH, Detemir or Glargine).
11. Subjects requiring other anti-diabetic medications other than insulin (oral or injectable).
12. Pregnancy
13. Sexually active females who do not practice acceptable contraceptive methods to prevent pregnancy.
14. Presence of a febrile illness within 24 hours of start ski camp or acetaminophen use while wearing the CGM. The camp study subject will not participate in the trial if these conditions are met.
15. Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

    * Inpatient psychiatric treatment in the past 6 months
    * Uncontrolled adrenal insufficiency
    * Alcohol abuse

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time in range when using closed-loop compared with SAP. | 120-144 hours

SECONDARY OUTCOMES:
Reduction of hypoglycemia episodes when using closed-loop | 120-144 hours
  assessed by the number of hypoglycemia treatments were needed for each group

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R. Chernavvsky, MD, CRC, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Colorado, Denver, Barbara Davis Center, Aurora, Colorado
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
undetermined

REFERENCES:
- [Result] Breton MD, Chernavvsky DR, Forlenza GP, DeBoer MD, Robic J, Wadwa RP, Messer LH, Kovatchev BP, Maahs DM. Closed-Loop Control During Intense Prolonged Outdoor Exercise in Adolescents With Type 1 Diabetes: The Artificial Pancreas Ski Study. Diabetes Care. 2017 Dec;40(12):1644-1650. doi: 10.2337/dc17-0883. Epub 2017 Aug 30. PMID 28855239